CLINICAL TRIAL: NCT06116201
Title: Influences of Long Term Hormone Therapy on Physical Fitness and Vascular Function in Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Prof. Dr.Daroonwan Suksom, Faculty of Sports Science, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SPSC-7
Record Dates: First submitted 2021-05-27; First posted 2023-11-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Transgender Women
Keywords: Transgender women; Physical fitness; Vascular function; Hormone therapy
MeSH Terms: interventions — Estradiol; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transgender women with orchiectomy (Experimental): Transgender women who took medication for sex transition form male to female via estradiol hormone therapy and orchiectomy surgery. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: Estradiol
- Transgender women without orchiectomy (Experimental): Transgender women who took medication for sex transition form male to female via estradiol hormone and anti-androgen hormone therapy. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: Estradiol and Anti-Androgen
- Cisgender men (Sham Comparator): Cisgender men who lived in normal life were not used medication process for sex transition. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: No intervention
- Cisgender women (Sham Comparator): Cisgender women who lived in normal life were not used medication process for sex transition. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Estradiol — Estradiol
  Arms: Transgender women with orchiectomy
Other: Estradiol and Anti-Androgen — Estradiol and Anti-Androgen
  Arms: Transgender women without orchiectomy
Other: No intervention — No intervention
  Arms: Cisgender men; Cisgender women

SUMMARY:
Transgender women who transitioned from male to female by hormone therapy demonstrate similar physical fitness and vascular function to males or females.

DETAILED DESCRIPTION:
This cross-sectional study was to compare physical fitness and vascular function between cisgender men, cisgender women, and transgender women.

ELIGIBILITY:
Inclusion Criteria:

1. Cisgender men group (Body mass index between 18.5-24.9 and NO NCDs).
2. Cisgender women group (Body mass index between 18.5-24.9, No pregnant, NO NCDs).
3. Transgender women with orchiectomy (Body mass index between 18.5-24.9, taking estradiol, testosterone level below 10 nmol/L, NO NCDs).
4. Transgender women without orchiectomy (Body mass index between 18.5-24.9, taking estradiol and anti-androgen, testosterone level below 10 nmol/L, NO NCDs).

Exclusion Criteria:

* Participants had an injury during testing.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men, Cisgender women, Transgender women with orchiectomy, Transgender women without orchiectomy
Enrollment: 60 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Heart rate | Baseline
  Heart rate will be measured with automated blood pressure device (CARESCAPE V100, GE Dinamap).
Blood pressure | Baseline
  Systolic blood pressure and diastolic blood pressure will be measured with automated blood pressure device (CARESCAPE V100, GE Dinamap). Mean arterial blood pressure was calculated from systolic blood pressure and diastolic blood pressure via mean arterial pressure formula.
Body weight | Baseline
  Body weight and height will be measured with automated body composition machine (ioi 353, Jawon medical).
Height | Baseline
  Height will be measured with automated body composition machine (ioi 353, Jawon medical).
Resting metabolic rate | Baseline
  Energy expenditure will be measured by canopy study protocol with stationary gas analyzer (VMAX, Encore 29 system).
Vascular structure | Baseline
  Intima-Media Thickness will be measured with ultrasonography equipment on carotid artery (EPIQ 5G, Phillips).
Macro vascular function | Baseline
  Macro vascular function will be measured by brachial artery flow-mediated dilatation protocol on brachial artery with ultrasonography equipment (EPIQ 5G, Phillips).
Arterial stiffness | Baseline
  Arterial stiffness will be measured with brachial-ankle pulse wave velocity (VP-1000 plus, omrom Healthcare).
Micro vascular function | Baseline
  Micro vascular function will be measured by post-occlusive hyperemia protocol of fingertip cutaneous blood flow with laser doppler flowmetry device (PeriFlux system 5000, Perimed).
Muscle mass | Baseline
  Muscle mass will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcaare).
Fat mass | Baseline
  Fat mass will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcaare).
Bone mineral content | Baseline
  Bone mineral content will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcaare).
Bone mineral density | Baseline
  Bone mineral density will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcaare).
T-score of bone density | Baseline
  T-score will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcaare). T-score was separated into 3 categories, 1 or higher of T-score that is the healthy bone, -1 to -2.5 of T-score that is osteopenia, and -2.5 or lower that is osteoporosis.
Cardiorespiratory fitness | Baseline
  Maximal oxygen consumption will be measured by Bruce protocol for treadmill test with stationary gas analyzer (VMAX, Encore 29 system).
Muscle strength and muscle endurance | Baseline
  Muscle strength and muscle endurance will be measured by concentric/concentric protocol with isokinetic machine (Biodex Multi-Joint System-Pro, Biodex).
Flexibility | Baseline
  Sit and reach test will be measured by sit and reach protocol with sit and reach box (Grandsport).
Agility | Baseline
  Agility will be measured by T-test protocol with timing gate device (SpeedLight Timing System, Swiftperformance).
Balance | Baseline
  Balance will be measured by balance error scoring system (BESS) protocol with postural sway detected machine (Biosway, Biodex).
Coordination and reaction time | Baseline
  Coordination and reaction time will be measured by eye-hand coordination protocol with light reacted device (FITLIGHT Trainer).
Muscular power | Baseline
  Muscular power will be measured by vertical jump with force plate detected machine (Ballistic Measurement System & FT 700 Power Cage, Fitness Technology).
Speed | Baseline
  Speed will be measured by sprint test for 40 meters with timing gate device (SpeedLight Timing System, Swiftperformance).
Anaerobic fitness | Baseline
  Anaerobic fitness will be measured by Wingate test protocol with ergocycle (Monark 894e).

SECONDARY OUTCOMES:
Quality of life level | Baseline
  Quality of life will level will be measured by World Health Organization Quality of Life Brief - Thai questionnaire. The scores of questionnaire were 130 points for maximum value and 26 points for minimum value. 3 levels in quality of life were less than 61 points for below normal range, 61-95 points for normal range, and more than 95 points for above normal range.
Stress level | Baseline
  Stress level will be measured by Suanprung Stress Test-20 questionnaire. The scores of questionnaire were 100 points for maximum value and 20 points for minimum value. 4 levels in stress less than 24 points for low stress range, 24-41 points for normal stress range, 42-61 points for high stress range, and more than 61 points for severe stress range.

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Study Director — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saitong A, Naeowong W, Suksom D, Tanaka H. Physical Fitness and Exercise Performance of Transgender Women. Med Sci Sports Exerc. 2025 Jan 1;57(1):134-143. doi: 10.1249/MSS.0000000000003536. Epub 2024 Aug 12. PMID 39140786